CLINICAL TRIAL: NCT07021638
Title: EMMVIES : Walking Training at Home in VIrtual Reality for Children With Chronic Illnesses Impacting Physical Health
Acronym: EMMVIES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 49RC24_0215; 2025-A01261-48 (Other: ANSM)
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Home-based Programs; EzyGain; AMY Treadmill; Cerebral Palsy; Neuromuscular Diseases (NMD); Obesity; Virtual Reality
MeSH Terms: conditions — Cerebral Palsy; Neuromuscular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMMVIES program (Experimental): Evaluate the feasibility of the home training program.
  Interventions: Other: EMMVIES program

INTERVENTIONS:
Other: EMMVIES program — Walking Training at Home in VIrtual Reality for Children with Chronic Illnesses Impacting Physical Health

SUMMARY:
Over the past 30 years, the prevalence of congenital or acquired chronic diseases in children has risen, affecting between 10 and 30% of them, or at least 100,000 children in France. Pathologies such as cerebral palsy (CP), neuromuscular diseases (NMD), obesity or congenital heart disease impact physical health by causing musculoskeletal, respiratory or cardiovascular deficiencies. These limitations influence their ability to participate in daily activities, affecting their quality of life and that of their families.To minimize these impacts, motor rehabilitation programs focusing on physical activity are proposed, but their effectiveness requires prolonged practice. However, these specific programs, often delivered in remote specialized centers, are difficult to access. Home programs have been developed to overcome these constraints. They enable children, with the support of their parents, to carry out therapeutic activities at home. Although their feasibility has been demonstrated, their effectiveness is relative. A multitude of protocols and tools have been tested, with no harmonization of practices.To support the implementation of home-based programs for children with CP or obesity, virtual reality has already been used, mainly on the basis of commercial solutions. This solution is therefore feasible and has proved relatively effective.With this in mind, and based on the user experience of children, parents and professionals, the investigators have initially co-developed with the French company EzyGain a connected treadmill specifically adapted to pediatric needs and the requirements of home programs. The AMY treadmill is a compact treadmill with on-board sensors and a safety system, communicating with a tablet application and a virtual reality headset.Taking into account the opportunities offered by this new technology, as well as building on the effects and features already known from home programs, the investigators have developed a new modality for home programs focusing on walking for children with CP, MNM and obesity, the EMMVIES program. The crucial step now is to investigate the feasibility, tolerance and clinical effects of this EMMVIES program.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 6 to 17 years at date of inclusion;
* Able to walk for 5 minutes on a treadmill with or without body weight support, with or without technical aids;
* Be able to understand and play virtual reality games (immersive or non-immersive);
* Be able to answer questionnaires;
* Patient affiliated to or benefiting from a social security scheme;
* Informed consent, dated and signed by parents or guardians (if minors), to participate in the study;
* Included in a care program specific to their chronic condition for at least 6 months;
* Meet the following criteria depending on the group:

PC group:

* Diagnosis of CP
* Functional level classified II or III according to the Gross Motor Function Classification System (GMFCS)
* Rehabilitation goal: improvement of gait and/or gross motor function

OB group:

* Overweight or obese, defined by a BMI above the IOTF-25 percentile
* Aim to increase daily physical activity
* No history of hip pathology

Group NM:

* Diagnosis of one of the following neuromuscular pathologies: spinal muscular atrophy type 3, Duchenne disease, congenital myopathy or Charcot Marie Tooth.
* Functional level of grade 2 to 6 on the Walton scale, or grade 3 to 7 on the Vignos scale
* Rehabilitation goal: improvement of walking and/or gross motor skills

Exclusion Criteria:

* Patients weighing over 100 kg (due to the technical constraints of using the AMY mat).
* For children aged 6 to 11: in connection with the immersive virtual reality device: problems with stereoscopic vision (perception of images in 3 dimensions), unstabilized epilepsy, facial trauma < 3 months, hearing or visual impairment, pain, dizziness or nausea caused by using immersive virtual reality.
* Patients who have undergone surgery in the last 3 months;
* Patients who have received intramuscular botulinum toxin injections in the lower limbs or intensive therapy in the 3 months prior to inclusion;
* Patient with a non-routine therapeutic program planned within 5 months that could lead to confusion with the tested program;
* Patient with insufficient understanding of the French language;
* Patient opposition (child or adolescent);
* Persons deprived of liberty by judicial or administrative decision;
* Persons under compulsory psychiatric care;
* Persons under legal protection;

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Home rehabilitation program | 3 x 30-minute sessions over 10 weeks
  The treadmill walking training program comprises a minimum of 3 sessions per week, with one day of rest between each session. Each session comprises around 30 minutes of physical exercise on a mat, alternating between walking and balance exercises.

SECONDARY OUTCOMES:
Assessment of lower limb muscle strength | Inclusion, 10 weeks and 20 weeks
  Muscle strength is measured using a wireless electronic hand dynamometer (DEM) (MicroFET 2) based on a standardized protocol used in clinical routine and performed on an examination table on the following muscle groups: plantar flexors (knee extended and flexed), knee flexors and extensors and hip abductors. The child is asked to contract each muscle group tested for 3 to 5 seconds, three times against the dynamometer held by an assessor. The average of the three peak pressures achieved for each muscle group tested is recorded. The estimated duration of these measurements is 15 minutes.
10-meter walk test | Inclusion, 10 weeks and 20 weeks
  Patients' gait quality is assessed using a minimal version of the Quantified Gait Analysis (QGA), which simply includes spatiotemporal, kinematic and electromyographic gait parameters. To this end, 10-meter barefoot walking tests at spontaneous (2 trials), fast (2 trials) and double-task speeds, i.e. walking and listing animal names (1 trial) and fruit names (1 trial), and finally with usual shoes and orthoses, are carried out. Walking tests are performed in comfortable clothing, as close to the body as possible, with uncovered legs (shorts). A walking frame is authorized for children who cannot walk 10 meters without one. The total duration of the assessment for the child is 20 minutes.
6-minute walk test | Inclusion, 10 weeks and 20 weeks
  Walking endurance is assessed by the 6-minute walking test (TDM6). According to the instructions for this test, the distance covered in 6 minutes is observed. Children are asked to walk as far as possible in 6 minutes on a 60-meter marked track in corridors. Children are fitted with shoes, orthoses and/or walking aids, depending on their habits. Footwear and technical aids must be identical between the 3 evaluation times T0, T1 and T2. An indication of the remaining test time is given to the children every minute by the investigator. The duration of the test for the child is estimated at 10 minutes.
Motion control assessment | Inclusion, 10 weeks and 20 weeks
  Somatosensory function is measured by the cortico-cinematic coherence (CKC) index, which reflects the correlation between electrical activity in the primary sensorimotor cortex (measured by conventional low-density electroencephalogram (EEG)) and displacement of the center of pressure (CoP) in standing static equilibrium for 2 minutes (measured by a force platform). This exploratory index will enable us to estimate the cortical processing of proprioceptive afferents in the lower limbs. The estimated duration of this measurement is 10 minutes.
Balance assessment | Inclusion, 10 weeks and 20 weeks
  Balance is assessed by 30-second unipodal hold tests (1 trial), if possible for the child, and 30-second bipodal hold tests under open-eye (1 trial), closed-eye (1 trial), foam (1 trial) and double-task conditions, i.e. counting backwards from 50 (1 trial). These tests are performed on a force platform (AMTI Accusway) to record the CoP's trajectory. The evaluation is scheduled to last 10 minutes.
Assessment of gross motor functions for children with CP | Inclusion, 10 weeks and 20 weeks
  The GMFM-66 is a 66-item quantitative observational scale for assessing gross motor function in children with cerebral palsy (CP). Five dimensions of gross motor function are tested: Dimension A: lying and rolling, Dimension B: sitting, Dimension C: crawling and kneeling, Dimension D: standing, Dimension E: walking, running and jumping. Each item is scored on a 4-point scale, depending on whether the task requested by the investigator has been completed in full or in part. A maximum of three trials is allowed, and any spontaneous performance is accepted. The GMFM 66 takes around 45 minutes to complete.
Assessment of gross motor functions for children with MNM | Inclusion, 10 weeks and 20 weeks
  For children with neuromuscular disorders (NMD), the Motor Function Measure (MFM). The MFM is a quantitative observational scale comprising 32 items, divided into 3 domains: domain D1: standing and transfer, domain D2: axial and proximal function, and domain D3: distal function. Each item assesses a specific motor task, and performance is rated on a scale from 0 to 3. The child is asked to perform the various MFM tasks. The MFM takes around 45 minutes to complete.
Quality of life assessment | Inclusion, 10 weeks and 20 weeks
  Quality of life is assessed by the KIDSCREEN questionnaire. The KIDSCREEN-27 measures health-related quality of life in children and adolescents aged 8 to 18, across five dimensions: physical well-being, psychological well-being, autonomy and relationships with parents, social support and relationships with peers, and school environment. In this study, only the dimensions of physical well-being, psychological well-being, autonomy and relationships with parents are assessed. The questionnaire is completed by the child, unless under 8 years of age. Approximate completion time for children is 5 minutes.
Assessment of daily activities and mobility | Inclusion, 10 weeks and 20 weeks
  Achievement of daily activities and mobility is assessed by the Pediatric Evaluation of Disability Inventory as a Computer Adaptive Test (PEDI-CAT). The PEDI-CAT measures the functional abilities of children with disabilities in four functional domains: activities of daily living, mobility, social and cognitive activities, and responsibility. The daily activities and mobility domains are assessed. The questionnaire is completed online during the consultation by the child accompanied by at least one parent. It takes approximately 15 minutes for the child to complete the questionnaire online.
Actimetry | Inclusion, 10 weeks and 20 weeks
  Daily physical activity (PA) is measured using an actimeter (Actigraph GT3X). The following parameters are observed: number of daily steps, time spent at different levels of phsyical activity intensity (sedentary, light, moderate to vigorous), and time spent in different positions (lying, sitting, standing). The actimeter is worn on a belt during the day and on the wrist at night, for 7 consecutive days before or after each visit.
User experience - User Experience Questionnaire | once at 20 weeks
  The short version of the User Experience Questionnaire (UEQ-S) is used. It contains 8 items grouped into two scales: pragmatic qualities (efficiency, insight, reliability) and hedonic qualities (stimulation, novelty). The format of the items is a semantic differential (e.g. Complicated - Simple) with a 7-point Likert scale. This questionnaire was chosen because it is the most widely used in the literature and has already been used with children.
User experience - Usability Metric for User Experience | once at 20 weeks
  The Usability Metric for User Experience (UMUX) is a short 4-item questionnaire. The items are statements about ease of use and usefulness, with which respondents express agreement on a 7-point Likert scale. The UMUX is strongly correlated with the System Usability Scale (SUS), which is the most widely used usability questionnaire, with a large amount of associated research literature, but contains 10 items. The scores obtained on the UMUX are therefore used to position the solution's usability on the SUS interpretation scale ("worst imaginable", "poor", "acceptable", "good", 'excellent' or "best imaginable").
User experience - Mobile Applications Rating Scale version utilisateur | once at 20 weeks
  The MARS (Mobile Applications Rating Scale user version) comprises 23 items divided into 6 domains. We will examine the first 3 domains: engagement, functionality and aesthetics. Answers are given on 5-point Likert scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Capucins, Angers, France

IPD SHARING:
Plan to Share IPD: No